CLINICAL TRIAL: NCT02212223
Title: Food-based Solutions for Optimal Vitamin D Nutrition and Health Through the Life Cycle (ODIN)
Brief Title: Marwo-D Research -Need for Vitamin D in Different Population Groups
Acronym: ODIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: University College Cork (Other); Technical University of Denmark (Other); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Christel Lamberg-Allardt, Associate Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Helsinki U
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Serum 25-hydroxyvitamin D Concentrations (25OHD)
Keywords: Vitamin D; Serum 25-hydroxyvitamin D (25OHD); Dietary supplement; Ethnicity; Immigrant
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1: Somali immigrant group, 10 µg (400 IU) vitamin D3 (Experimental): Subjects belonging to Somali immigrant population are given a daily supplement containing 10 µg (400 IU) vitamin D3 to take for 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Group 2: Somali immigrant group, 20 µg (800 IU) vitamin D3 (Experimental): Subjects belonging to Somali immigrant population are given a daily supplement containing 20 µg (800 IU) vitamin D3 to take for 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Group 3: Somali immigrant group, 0 µg vitamin D3 (Placebo Comparator): Subjects belonging to Somali immigrant population are given a daily supplement containing 0 µg (0 IU) vitamin D3 to take for 6 months
- Group 4: Original Finnish group, 10 µg (400 IU) vitamin D3 (Experimental): Subjects belonging to original Finnish population are given a daily supplement containing 10 µg (400 IU) vitamin D3 to take for 6 months.
  Interventions: Dietary Supplement: Vitamin D3
- Group 5: Original Finnish group, 20 µg (800 IU) vitamin D3 (Experimental): Subjects belonging to original Finnish population are given a daily supplement containing 20 µg (800 IU) vitamin D3 to take for 6 months.
  Interventions: Dietary Supplement: Vitamin D3
- Group 6: Original Finnish group, 0 µg vitamin D3 (Placebo Comparator): Subjects belonging to original Finnish population are given a daily supplement containing 0 µg (0 IU) vitamin D3 to take for 6 months.

INTERVENTIONS:
Dietary Supplement: Vitamin D3
  Arms: Group 1: Somali immigrant group, 10 µg (400 IU) vitamin D3; Group 2: Somali immigrant group, 20 µg (800 IU) vitamin D3; Group 4: Original Finnish group, 10 µg (400 IU) vitamin D3; Group 5: Original Finnish group, 20 µg (800 IU) vitamin D3

SUMMARY:
Insufficient intake of vitamin D is a public health problem, affecting about 40% of the Finnish population in the winter. Vitamin D has a wide range of health effects: in addition to its effect on bone, it is known to affect inflammatory response among other things. The sources of vitamin D are the synthesis in the skin as well as diet and dietary supplements. In Finland and in Northern Europe vitamin D is formed in the skin only from March to October. This alone is not sufficient to cover the need for year-round, because vitamin D storage is used in a few months. During the winter months the only sources of vitamin D are diet and vitamin preparations. Current vitamin D recommendations are usually based on studies in white population. However, there can be a difference in the need of vitamin D and in vitamin D metabolism between different population groups. More research evidence is needed from the northern countries. The aim of this study is to evaluate the vitamin D need in Somali immigrant population and in original Finnish population. The hypothesis is that the Somalis need more vitamin D to exceed the serum 25(OH)D concentration of 50 nmol/L than the original Finnish population.

ELIGIBILITY:
Inclusion Criteria:

* woman between 21-66 years of age
* belongs to original Finnish population or to Somali immigrant population
* healthy (= no disease requiring medication)
* lives in the metropolitan area

Exclusion Criteria:

* pregnant or breastfeeding
* has traveled to a sunny destination or destination near the equator during the previous month
* plans to travel to a sunny destination or destination near the equator in the next 6 months
* has used a tanning bed during the previous month
* plans to use a tanning bed in the next 6 months
* the subject's blood 25-hydroxy-vitamin D level (25 (OH) D), exceeds 100 nmol / L or is less than 30 nmol / L at baseline in the screening phase.

Ages: 21 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D (25(OH)D) concentrations | Change from baseline in serum 25(OH)D concentration at 3 and 6 months
  The effect of ethnicity on the serum 25(OH)D concentration response to vitamin D supplementation will be investigated.

SECONDARY OUTCOMES:
Serum calcium concentration | Change from baseline in serum calcium concentration at 3 and 6 months
  Markers of calcium metabolism, which are affected by vitamin D, will be measured
Serum parathyroid hormone (PTH) concentration | Change from baseline in serum PTH concentration at 3 and 6 months
  Markers of calcium metabolism, which are affected by vitamin D, will be measured

OTHER OUTCOMES:
Polymorphisms in genes involved in the transport and metabolism of vitamin D | Baseline
  Genomic DNA will be isolated and single nucleotide polymorphisms (SNPs) for key genes involved in vitamin D transport and metabolism will be measured to investigate the ethnic variation in the genes.

CONTACTS AND LOCATIONS:
Overall Officials: Christel Lamberg-Allardt, Professor, Study Director — University of Helsinki
Locations (1):
- Department of Food and Environmental Sciences, University of Helsinki, Helsinki, Finland